CLINICAL TRIAL: NCT06352359
Title: Safety, Pharmacokinetics (PK), and Efficacy of ONC 841 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-841-002
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONC-841 (Experimental): ONC-841 will be given by IV infusion in designated dose, q4w.
  Interventions: Drug: ONC-841

INTERVENTIONS:
Drug: ONC-841 — ONC-841 (anti-SIGLEC10) is a humanized antibody that binds to human sialic acid-binding Ig-like lectin 10 and has a human immunoglobulin G4 (IgG4) Fc domain.
  Other Names: Anti-SIGLEC10 antibody

SUMMARY:
This is a Phase I open label, dose-escalation study of intravenous (IV) infusion of ONC-841 as a single agent in patients with advanced/metastatic solid tumors. The study will evaluate seven dose levels of ONC-841 starting from 0.03 mg/kg to 30 mg/kg.

DETAILED DESCRIPTION:
ONC-841 is an investigational drug being developed as an anti-tumor treatment. ONC-841 is an antibody drug that binds to immune cells inside the tumor mass. The target molecule is Siglec10, mostly expressed on neutrophils, macrophages and lymphocytes. ONC-841 binds to Siglec10 to block the "do not eat me" signals that cancer cells give to immune system, which allow macrophages and neutrophils to "eat" the tumor cells. The study will use ONC-841 alone for cancer treatment. The study will evaluate seven dose levels of ONC-841 starting from 0.03 mg/kg to 30 mg/kg, given once every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have ECOG score ≤ 1. The body weight should be ≥40 kg.
* A histological or cytological diagnosis of solid tumors and metastatic disease or locally advanced disease.
* Must have measurable target lesion according to RECIST V1.1.
* Adequate organ function as determined by laboratory tests.
* Voluntary agreement to participate as evidenced by written informed consent.
* Female patient: negative pregnancy test and agreement on contraceptive methods.
* Male patient: agreement on contraceptive methods.
* Agree to give archival or other diagnostic tissue recut slides or an optional new tumor biopsy.

Exclusion Criteria:

* Patients who have not recovered to NCI CTCAE grade ≤ 1 from an adverse event (AE) due to cancer therapeutics except the chemotherapy-associated peripheral neuropathy (motor or sensory) or alopecia. Patients with ongoing and adequately controlled endocrine immune-related AEs are considered stable and eligible for enrollment.
* The washout period for cancer therapeutic drugs should be 5 half-life or 21 days for chemotherapy, whichever is shorter; or 28 days for monoclonal antibody therapy. Palliative radiotherapy for painful metastases or metastases in potentially sensitive locations (e.g., epidural space) ≥ 7 days prior to the first dose of study drug. Best supportive care, such as thyroxine, insulin, steroid replacement treatment, blood transfusion and therapy for non-cancer conditions are allowed.
* Patients who are currently enrolled in any other clinical trial testing an investigational agent or device, or with concurrent anticancer treatment (except palliative bone-directed radiotherapy), immune therapy, or cytokine therapy or anticipated to require another antineoplastic therapy during the study.
* Patients who are on chronic systemic steroid therapy at doses higher than 10 mg/day prednisone or equivalent within 7 days before first treatment.
* Patients who have active brain metastases or leptomeningeal metastases. Patients who have active brain metastases or leptomeningeal metastases. Patients are eligible if brain metastases are adequately treated, and patients are asymptomatic or neurologically stable (except for residual signs or symptoms related to the central nervous system (CNS) treatment). Note: Patients with previously treated brain metastases may participate provided they are radiologically stable (i.e. no evidence of progression for ≥4 weeks by repeat imaging performed during study screening), clinically stable, and not requiring steroid treatment within 14 days before the first dose of study treatment.
* Patient with a different cancer other than the one treated under this protocol, which requires systemic treatments within 24 months prior to C1D1.
* Patient has history of grade ≥3 allergic or hypersensitivity to IV infusion medications, or severe allergic reactions to food, pollen, oral medications, or atopic dermatitis or asthmatic episodes that required hospitalization.
* Within past 6 months with history of significant cardiovascular acute myocardial infarction, acute coronary syndrome, ischemic or hemorrhagic stroke, revascularization procedures, acute pulmonary embolism or any disorders resulted in LVEF < 40% at the time of screening or colitis, small bowel obstruction, hepatitis or pancreatitis adrenal insufficiency, or severe immunotherapy related AE (irAE≥ grade 3).
* Patients who have acute infections which require systemic treatments within 14 days prior to C1D1.
* Patients who, in the opinion of the treating Investigator, have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or make study participation not in the best interest of the patient, in the opinion of the treating Investigator. Investigators should discuss the case with the Sponsor and/or study leaders.
* Patients with known psychiatric or substance abuse disorders may interfere with cooperation with the requirements of the trial.
* Patients who are pregnant or breastfeeding or plan pregnancy or fathering the child during the study or within 6 months after the last dosing of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 28 Days
  The number of subjects who have Dose limiting toxicity (DLT) as defined by protocol DLT criteria during the first cycle of study drug, ONC-841, administration.
Maximum Toxicity Dose (MTD) | 28 Days
  Maximal tolerable dose (MTD), the study drug, ONC-841, dose level that has two out of six subjects who have DLT.

SECONDARY OUTCOMES:
Cmax of ONC-841 | 84 days
  The highest Serum concentration of ONC-841 after IV infusion at cycle 1 and cycle 3 from different timepoints (within 60 minutes before dosing, 60 minutes post-dose, 6 hours post-dose, 24 hours post dose, day 8, 15 and 21 post-dose) after drug administration.
The serum half-life of ONC-841 | 84 days
  To determine the drug concentration in serum samples that are taken in various timepoints (Cycle 1 and Cycle 3: within 60 minutes before dosing, 60 minutes post-dose, 6 hours post-dose, 24 hours post dose, day 8, 15 and 21 post-dose. Cycle 2 and Cycle 4-13: within 60 minutes before dosing and 60 minutes post-dose) during the treatment in order to calculate drug half life.

CONTACTS AND LOCATIONS:
Overall Officials: Tianhong Li, MD, PhD, Principal Investigator — University of California, Davis
Locations (8):
- United States (8):
  - University of California at Davis Cancer Center, Sacramento, California
  - UF Health Cancer Center, University of Florida, Gainesville, Florida
  - AdventHealth Medical Group Oncology Research at Celebration, Kissimmee, Florida
  - Norton Cancer Center, Louisville, Kentucky
  - Rogel Cancer Center, University of Michigan, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - Tranquil Clinical Research, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No